CLINICAL TRIAL: NCT01121926
Title: A Randomized, Two-way Crossover Study to Compare the Bioavailability of 300 mg Trazodone Hydrochloride Extended-release Caplets (Containing Contramid®) (Administered Once Daily) and 100 mg Trazodone Hydrochloride Immediate-release Tablets (Administered Three Times Daily) at Steady State
Brief Title: A Study to Compare the Bioavailability of 300 mg Trazodone Hydrochloride Extended-release Caplets and 100 mg Trazodone Hydrochloride Immediate-release Tablets at Steady State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 04ACL108
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2010-08-16 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Subjects; Bioavailability; Pharmacokinetics
Keywords: Healthy subjects; Bioavailability; Pharmacokinetics; Trazodone; Steady-state
MeSH Terms: interventions — Trazodone

ARMS (2):
- Trazodone HCl OAD (Experimental): OAD: Once A Day
  Interventions: Drug: Trazodone HCl
- Trazodone HCl (Apotex Corp.) (Active Comparator)
  Interventions: Drug: Trazodone HCl

INTERVENTIONS:
Drug: Trazodone HCl — Dosage form:
  Extended-release caplets containing 300 mg trazodone HCl and extended-release caplets containing 150 mg trazodone HCl (the 150 mg dosage form was only used for the up and down titration, and was not evaluated in the study).
  Dose regimen:
  75 mg trazodone HCl (½ x 150 mg extended-release caplet) on Days 1 and 11, 150 mg trazodone HCl (one extended-release caplet) on Days 2 and 10, 300 mg trazodone HCl (one extended-release caplet) on Days 3 to 9, each at 23:30 after a fast of at least 4 hours.
  Other Names: Oleptro
  Arms: Trazodone HCl OAD
Drug: Trazodone HCl — Dosage form:
  Immediate-release tablet containing 100 mg trazodone HCl
  Dose regimen:
  100 mg trazodone HCl (one immediate-release tablet) once (at 23:30) on Days 1 and 11, 100 mg trazodone HCl (one immediate-release tablet) twice (at 23:30 and 11:30) on Days 2 and 10, 100 mg trazodone HCl (one immediate-release tablet) three times daily (at 23:30, 07:30 and 15:30) on Days 3 to 9. Evening doses were administered after a fast of at least 4 hours.
  Arms: Trazodone HCl (Apotex Corp.)

SUMMARY:
The purpose of this study was to compare the pharmacokinetic profiles at steady state of the test product, 300 mg trazodone hydrochloride (HCl) extended-release caplets (containing Contramid®), when administered once daily, and the reference product, 100 mg trazodone HCl immediate-release tablets (Apotex Corp.), when administered three times daily, for one week. For this purpose, the rate and extent of absorption of trazodone and formation of m-chlorophenylpiperazine (mCPP) after administration of multiple doses of up to 300 mg of each of the two formulations was compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects 18 to <56 years of age.
* Body mass within 10% of ideal mass in relation to height and age, according to Body Mass Index.
* Body mass not less than 60 kg.
* Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results within the reference ranges for the relevant laboratory tests (unless the investigator considered the deviation to be irrelevant for the purpose of the study).
* Normal electrocardiogram (ECG) and vital signs, or abnormalities which the investigator did not consider a disqualification for participation in the study.
* Willingness to undergo pre- and post-study physical examinations and laboratory investigations.
* Ability to comprehend and willingness to sign both statements of informed consent (for screening and phase-related procedures).
* Non-smoker or past smoker who stopped the use of any form of tobacco, including snuff or similar products, at least 3 months before entering the study.
* For females, the following conditions had to be met:

  1. had been surgically sterilized or undergone a hysterectomy, or
  2. was of childbearing potential, and all of the following conditions were met:

     1. Had a negative pregnancy test at screening. If this test was positive, the subject was to be excluded from the study before receiving study medication. In the circumstance that a pregnancy was discovered after the subjects received the study medication, every attempt had to be made to follow such subjects to term.
     2. Had to agree to use an accepted method of contraception (i.e., spermicide and barrier methods or spermicide and non-hormonal intrauterine contraceptive device). The subject had to agree to continue with the same method throughout the study. Hormonal contraceptives were not allowed.
  3. females not of childbearing potential could also have been included if they had no menstrual period for one year and were considered as post-menopausal.

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* History of, or current compulsive alcohol abuse (>10 drinks weekly), or regular exposure to other substances of abuse.
* Use of any medication, prescribed or over-the-counter, within 2 weeks prior to the first administration of study medication except if this would not affect the outcome of the study in the opinion of the investigator.
* Participation in another study with an experimental drug, where the last administration (of previous study medication) was within 8 weeks before the first administration of study medication.
* Treatment within the previous 3 months with any drug with a well-defined potential for adversely affecting a major organ or system with evidence to this effect.
* A major illness during the 3 months before commencement of the screening period.
* History of hypersensitivity to the study medication or any related medication.
* History of bronchial asthma.
* History of epilepsy.
* History of porphyria.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
* Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of study medication.
* Diagnosis of hypotension made during the screening period.
* Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
* Resting pulse of > 100 beats per minute or < 40 beats per minute during the screening period, either supine or standing.
* Positive testing for HIV and/or Hepatitis B and/or Hepatitis C.
* Positive urine screen for drugs of abuse.
* Positive urine screen for tobacco use.
* A serum pregnancy test (beta human chorionic gonadotropin [β-HCG]) either positive or not performed or lactation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

REFERENCES:
- See also: Approved labelling — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=17925

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Trazodone Contramid® OAD) First: Trazodone Contramid® OAD (Once-A-Day) test product (300 mg tablet administered once daily) dosed in first treatment phase followed by Trazodone IR (Apotex Corp.) reference product (100 mg tablet administered thrice daily) dosed in the second treatment phase. A drug-free period of 7 calendar days separated the last administration of study medication in Phase 1 and the first administration of study medication in Phase 2.
  IR = Immediate Release.
- Reference (Trazodone IR [Apotex Corp.]) First: Trazodone IR (Apotex Corp.) reference product (100 mg tablet administered thrice daily) dosed in first treatment phase followed by Trazodone Contramid® OAD (Once-A-Day) test product (300 mg tablet administered once daily) dosed in the second treatment phase. A drug-free period of 7 calendar days separated the last administration of study medication in Phase 1 and the first administration of study medication in Phase 2.
  IR = Immediate Release.
Period: First Intervention Period
Arm/Group | Test (Trazodone Contramid® OAD) First | Reference (Trazodone IR [Apotex Corp.]) First
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout Period
Arm/Group | Test (Trazodone Contramid® OAD) First | Reference (Trazodone IR [Apotex Corp.]) First
Started | 14 | 15
Completed | 14 | 13
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Positive pregnancy test | 0 | 1
Period: Second Intervention Period
Arm/Group | Test (Trazodone Contramid® OAD) First | Reference (Trazodone IR [Apotex Corp.]) First
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Trazodone Contramid® OAD (Once-A-Day) test product first and Trazodone IR (Apotex Corp.) reference product first.
  IR = Immediate Release
Arm/Group | Entire Study Population
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Region of Enrollment [Number; unit: participants]
  South Africa | 30

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence Based on Cmax,ss
Description: Cmax,ss = Maximum plasma concentration (Cmax) at steady state (ss): (Cmax,ss). Measured in nanograms per milliliter (ng/mL).
Time Frame: 9 days
Population: The dataset for pharmacokinetic analysis comprised the 27 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Trazodone Contramid® OAD: Trazodone Contramid® OAD test product (300 mg tablet administered once daily) dosed in either period. A drug-free period of 7 calendar days separated the last administration of study medication in Phase 1 and the first administration of study medication in Phase 2.
- Trazodone HCl (Apotex Corp.): Trazodone HCl (Apotex Corp.) reference product (100 mg tablet administered thrice daily) dosed in either period. A drug-free period of 7 calendar days separated the last administration of study medication in Phase 1 and the first administration of study medication in Phase 2.
Arm/Group | Trazodone Contramid® OAD | Trazodone HCl (Apotex Corp.)
Number analyzed (Participants) | 27 | 27
ng/mL | 1812.026 (620.625) | 3117.778 (757.508)
Statistical Analysis 1: Comparison: Trazodone Contramid® OAD vs Trazodone HCl (Apotex Corp.); Test type: Non-Inferiority or Equivalence — Bioequivalence is established when the ratio of geometric Least Squares means (LSmeans) and confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter Cmax,ss is between 80% and 125%; Mean ratio = 56.53, 90% CI 2-sided [49.99 to 63.94] — Test/reference (%)

2. Primary Outcome: Bioequivalence Based on AUCss
Description: AUCss = Area under the plasma concentration curve (AUC) vs. time data pairs at steady state (ss): AUCss.
  Measured in nanograms x hours per milliliter (ng*h/mL).
Time Frame: 9 days
Population: The dataset for pharmacokinetic analysis comprised the 27 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Trazodone Contramid® OAD | Trazodone HCl (Apotex Corp.)
Number analyzed (Participants) | 27 | 27
ng*h/mL | 29131.374 (9930.767) | 33058.024 (8006.118)
Statistical Analysis 1: Comparison: Trazodone Contramid® OAD vs Trazodone HCl (Apotex Corp.); Test type: Non-Inferiority or Equivalence — Bioequivalence is established when the ratio of geometric Least Squares means (LSmeans) and confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter AUCss is between 80% and 125%; Mean ratio = 85.72, 90% CI 2-sided [81.05 to 90.67] — Test/reference (%)

3. Secondary Outcome: Minimum Plasma Concentration (Cmin,ss)
Description: Minimum plasma concentration at steady state (Cmin,ss). Measured in nanograms per milliliter (ng/mL)
Time Frame: 9 days
Population: The dataset for pharmacokinetic analysis comprised the 27 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Trazodone Contramid® OAD | Trazodone HCl (Apotex Corp.)
Number analyzed (Participants) | 27 | 27
ng/mL | 673.889 (354.647) | 842.763 (273.592)

4. Secondary Outcome: Plasma Concentration at 24 Hours Post-evening Dose (C24h)
Description: Plasma concentration at 24 hours post-evening dose (C24h) in nanograms per milliliter (ng/mL)
Time Frame: 9 days
Population: The dataset for pharmacokinetic analysis comprised the 27 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Trazodone Contramid® OAD | Trazodone HCl (Apotex Corp.)
Number analyzed (Participants) | 27 | 27
ng/mL | 747.270 (329.025) | 919.111 (289.382)

5. Secondary Outcome: Time to Peak Exposure (Tmax)
Description: Time to peak exposure (Tmax) at steady state.
Time Frame: 9 days
Population: The dataset for pharmacokinetic analysis comprised the 27 subjects who completed the study as per protocol.
Measure: Median (Full Range); unit: hours
Arm/Group | Trazodone Contramid® OAD | Trazodone HCl (Apotex Corp.)
Number analyzed (Participants) | 27 | 27
hours | 8.00 [3.00 to 16.0] | 8.33 [8.33 to 19.0]

6. Secondary Outcome: Percentage Swing
Description: Percentage swing is a pharmacokinetic parameter calculated as follows:
  ((Cmax,ss - Cmin,ss)/Cmin,ss)*100.
  Where:
  Cmax,ss = Maximum concentration at steady state; Cmin,ss = Minimum concentration at steady state.
  It was calculated over 24 hours on day 9.
Time Frame: 9 days
Population: The dataset for pharmacokinetic analysis comprised the 27 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: Percentage swing
Arm/Group | Trazodone Contramid® OAD | Trazodone HCl (Apotex Corp.)
Number analyzed (Participants) | 27 | 27
Percentage swing | 210.769 (127.806) | 302.805 (144.467)

7. Secondary Outcome: Percentage Peak-Trough Fluctuation (%PTF)
Description: Percentage Peak-Trough Fluctuation (%PTF) of trazodone calculated as [100*(Cmax-Cmin)/Cav].
  Cmax: Maximum plasma concentration Cmin: Minimum plasma concentration Cav: Average plasma concentration
Time Frame: 9 days
Population: The dataset for pharmacokinetic analysis comprised the 27 subjects who completed the study as per protocol.
Measure: Mean (Standard Deviation); unit: Percentage Peak-Trough Fluctuation
Arm/Group | Trazodone Contramid® OAD | Trazodone HCl (Apotex Corp.)
Number analyzed (Participants) | 27 | 27
Percentage Peak-Trough Fluctuation | 97.090 (28.357) | 174.768 (69.648)

ADVERSE EVENTS:
Arm/Group | Trazodone Contramid® OAD | Trazodone HCl (Apotex Corp.)
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 11/28 | 13/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trazodone Contramid® OAD (N=28) | Trazodone HCl (Apotex Corp.) (N=29)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Dizziness (Nervous system disorders) | 2 (3) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication based on the results of this study is envisaged, approval from the Sponsor will be obtained and a draft manuscript will be submitted to the sponsor for scrutiny and comment. The choice of scientific journal will be mutually agreed on by the principal investigator and the sponsor.